CLINICAL TRIAL: NCT01659047
Title: A Phase 2, Single-Arm, Open-Label Study Evaluating the Efficacy and Safety of Single Agent GS 1101 (CAL 101) as Therapy for Previously Treated Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-312-0120
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; CAL-101; Ofatumumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GS-1101 (Experimental): GS-1101 (oral; 150 mg BID)
  Interventions: Drug: GS-1101

INTERVENTIONS:
Drug: GS-1101 — 150 mg taken twice daily by mouth
  Other Names: CAL-101

SUMMARY:
The purpose of this study is to evaluate the effect of GS-1101 on the onset, magnitude, and duration of tumor control

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, single-arm, controlled, clinical trial evaluating the efficacy and safety of the phosphatidylinositol 3-kinase delta (PI3K-delta) inhibitor GS-1101 (CAL-101) as therapy for previously treated chronic lymphocytic leukemia.

This clinical trial (Study GS-US-312-0120) is a single-arm in which compliant subjects from GS US-312-0119 -Arm B who experience progression of CLL while receiving single-agent ofatumumab therapy are potentially eligible to receive single-agent, open-label GS 1101 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Study GS-US-312-0119
* Occurrence of confirmed progression of CLL while receiving single-agent ofatumumab in Study GS US 312 0119.
* Permanent cessation of Study GS-US-312-0119 (single-agent ofatumumab) and no intervening or continuing therapy (including radiotherapy, chemotherapy, immunotherapy, or investigational therapy) for the treatment of CLL.
* The time from permanent cessation of single-agent ofatumumab on Study GS-US-312-0119 and the initiation of GS 1101 on Study GS-US-312-0120 is no more than 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 18 mon
Patient Well-Being | 18 months
  Health-related quality-of-life questionnaire
Disease-related Biomarkers | 18 months
Pharmacokinetics | 6 months
  Evaluation of plasma concentrations at peak (Cmax) and trough (Cmin)
Incidence of Adverse Events | 18 months
Health Resource Utilization | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Langdon Miller, MD, Study Director — Gilead Sciences